CLINICAL TRIAL: NCT02234349
Title: Impact of Duodena-pancreatic Transplantation on Bile Acids and Incretins Metabolism.
Brief Title: Bile Acids and Incretins in Pancreas Kidney Transplant Patients
Acronym: ITABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012.768; 2012-A01517-36 (Registry Identifier: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Pancreas-kidney Transplantation; Kidney Transplantation
Keywords: bile acids; pancreas kidney transplantation; incretins; intestinal flora
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pancreas kidney transplant (Experimental): Patients with pancreas kidney transplantation
  Interventions: Procedure: pancreas kidney transplantation
- kidney transplant subjects (Experimental): Patients with kidney transplantation
  Interventions: Procedure: kidney transplantation
- Control (No Intervention)

INTERVENTIONS:
Procedure: pancreas kidney transplantation
  Arms: pancreas kidney transplant
Procedure: kidney transplantation
  Arms: kidney transplant subjects

SUMMARY:
Pancreas Kidney Transplantation (PKT) is the prominent treatment for type 1 diabetic patients with chronic kidney disease and improves patients' outcome. However, in spite of an optimized systemic insulin substitution, altered glucose metabolism and beta cell function are reported in these patients. The mechanisms behind these abnormalities are still unclear. Duodena-pancreatic anastomosis is performed in a heterotopic site (ileum) and thus could change physical and chemical properties of intestinal secretions, gut flora, as well as intestinal permeability. The effect of this procedure on gut derived metabolic factors, the enterohepatic cycle of bile acids, incretin secretion and intestinal flora have never been studied. This pilot prospective, study is aimed to evaluate the modification of bile acids concentrations and composition in PKT subjects, and the impact in glucose and incretin metabolism (measured by oral glucose tolerance test) one year after transplantation. The results will be compared to those of kidney transplant patients and control subjects.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* BMI <30 kg/m2
* Candidate for a first kidney transplant with a donor without the United Network for Organ Sharing (UNOS) criteria of extended donors and including living donors and pancreas-kidney donors (duodena-pancreas with ileal anastomosis and systemic drainage)
* Patients with conventional immunosuppression (maintenance with steroids, Tacrolimus and Mycophenolate Mofetil
* Willing and able to give informed consent

Control subjects :

* Potential living kidney donor

Exclusion Criteria:

* Subjects with a history of colectomy, gut resection or cholecystectomy
* For women : pregnancy
* Type 2 diabetes
* Type 1 diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Bile acids concentrations | One year after transplantation
  Plasmatic bile acids concentration will be measured in serum by biochemical analysis
Bile acids composition | One year after transplantation
  Plasmatic bile acids composition will be assessed in serum by gas chromatography

SECONDARY OUTCOMES:
Relationship between bile acid modifications and Oral Glucose Tolerance test (OGT) measures | One year after transplantation
  OGT will be performed in all subjects. Data on insulin sensitivity and secretion, Glucagon-Like Peptide 1 (GLP-1) and fibroblast growth factor-19 will be collected
Impact of Pancreas-Kidney Transplantation (PKT) on LipoPolySaccharides (LPS) | One year after transplantation
  LPS level will be measured before transplantation and one year after transplantation
Impact of PKT on intestinal flora | One year
  Gut microbiota will be analysed before and after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MORELON, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edourad Herriot - Pavillon P, Lyon, France

REFERENCES:
- [Result] Fitsum Guebre-Egziabher, Pascaline Alix, Charlotte Brunelle, Christophe Sulage ROLE OF BILE ACIDS IN NEPHROTIC SYNDROME ASSOCIATED DYSLIPIDEMIA Nephrology Dialysis Transplantation, Volume 32, Issue suppl_3, May 2017, Page iii589